CLINICAL TRIAL: NCT01899924
Title: Cognitive Assessment of Patients With Brain Injuries by the Mean of Event
Brief Title: Cognitive Assessment by the Mean of Event Related Potentials
Acronym: PEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I12011
Record Dates: First submitted 2013-06-27; First posted 2013-07-16 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Event Related Potentials (Experimental)
  Interventions: Behavioral: Event Related Potentials recording

INTERVENTIONS:
Behavioral: Event Related Potentials recording

SUMMARY:
The main objective of this study is to describe differential cognitive processing of various stimuli by a population of control subjects and a population of patients with selective cognitive deficits or altered states of consciousness by using dedicated ERP paradigms and high-density EEG picked up system.

DETAILED DESCRIPTION:
In order to test the relevance of theoretical models of cognitive functions, examination of patients with cerebral lesions is of great interest. Thus, the goal of this study is to assess cognitive processing in patients by a combination of behavioural clinical tests and ERP (event related potentials) specific markers. Indeed, ERP technique makes it possible to ascertain that a patient or control subject has or has not performed the task we asked him to even if the subject performs the task covertly. From these ERPs markers, we can investigate their respective cortical generators. By comparing the results obtained in both healthy and pathological populations, we will be able to appreciate differential processing of the same stimuli by two different populations and try to correlate these differences with specific cerebral lesions and with different outcomes.We previously demonstrated the relevance of this approach in the field of disorders of consciousness patients and we project to enrich this specific approach by the addition of new markers and by its extension to other fields of cognitive and behavioural neurology.

The procedure will be the following. After obtaining written informed consent, patients will be examined clinically with dedicated specialized scales (for example the CRS-R for disorders of consciousness patients). Then, we will probe event related potentials by stimulating these patients with various stimuli embedded in well-designed paradigms while their scalp EEG will be recorded. Following different steps of signal processing the mean ERPs according to conditions will be extracted and statistical analysis will be performed. At one year from the recording, outcome will be collected and correlated with the obtained ERPs.

ELIGIBILITY:
Control subjects

Inclusion Criteria:

* adults between 18 and 80,
* written informed consent obtained from the subject,
* covers by social insurance,
* absence of psychoactive drug intake in the week preceding the examination or alcohol intake the day before the exam

Exclusion Criteria:

* pregnant patients or breastfeeding,
* sensory deficit incompatible with the participation in tne study,
* person under a legal protection measure, under guardianship,
* psychoactive drug intake in the week preceding the examination or alcohol intake the day before the exam

Patients :

Inclusion Criteria:

* adults between 18 and 80,
* written informed consent obtained from the patient or his relatives,
* covers by social insurance,
* patients with either focal or diffuse brain damage drom trauma, vascular, tumor or other aetiologies, or with a history of neonatal or congenital diseases,
* patients with selective cognitive disorders or with altered states of consciousness

Exclusion Criteria:

* Pregnant patients or breastfeeding,
* sensory deficit incompatible with the participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2013-07; Primary Completion 2017-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Cognitive processing assessment | Day1
  Specific Event Related Potential (ERP) presence. ERP measurements indicate if a patient or control subject has or has not performed the task we asked him to even if the subject performs the task covertly

SECONDARY OUTCOMES:
Scalp topographies of ERPs | Day 1
  Links between the performance of a given task and the brain areas cognitive function.
Cognitive assessment by means of specialized scales | Day1, Day 356
  Patients will be examined clinically with dedicated specialized scales:
  CRS-R (Coma Recovery Scale- Revised), GOSE (Glasgow Outcome Scale Extended) and other dedicated scorings.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU of Limoges, Limoges, France